CLINICAL TRIAL: NCT05467748
Title: Phase Ib/II Study of Safety and Efficacy of EZH2 Inhibitor, Tulmimetostat, and PD-1 Blockade for Treatment of Advanced Non-small Cell Lung Cancer
Brief Title: EZH2 Inhibitor, Tulmimetostat, and PD-1 Blockade for Treatment of Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPLP-002-21F; 1673664 (Other: Michael E. Debakey VA Medical Center)
Record Dates: First submitted 2022-07-13; First posted 2022-07-20 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: PD-1 blockade; EZH2 inhibitor; Immunotherapy; Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase IB: Determine RP2D of tulmimetostat by using BOIN design with 2 dose levels, 200 and 300 mg once daily in combination of standard pembrolizumab 200 mg IV every 3 weeks. Tulmimetostat is currently under evaluation as single agent for patients with various solid tumors.
  Phase II: Based on Simon Optimum two stage design, our total number of patients for phase II is 54 patients (patients treated with RP2D from phase IB will be included in the analysis). We will enroll 15 patients at first stage to determine futility of the trial and complete the remaining 39 patients during stage II.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- combination of tulmimetostat and pembrolizumab (Experimental): Enrolled patients will receive combination treatment for whole study duration (2 years). For first cycle, patient will start tulmimetostat one week prior to start every 3 week pembrolizumab intravenous infusion (pembrolizumab will be given day 8 only for the first cycle, rest of cycles will be day 1 of each cycle).
  Interventions: Drug: Tulmimetostat

INTERVENTIONS:
Drug: Tulmimetostat — combination of oral tazemetostat and intravenous pembrolizumab treatment for patients with advanced non-small cell lung cancer
  Other Names: Pembrolizumab

SUMMARY:
This is an open label, single arm, phase Ib/II clinical trial of checkpoint blockade, pembrolizumab and EZH2 inhibitor, tulmimetostat combination therapy for patients with advanced non-small cell lung cancer who have progressed from front or second-line treatment. Patients will be enrolled at multiple Veterans Affairs Medical Centers.

DETAILED DESCRIPTION:
It is pleasing to witness the fulfillment of the promise of cancer immunotherapy becoming a reality for patients with many types of advanced cancer. However, even with this remarkable progress, majority of patients are not responding and substantial number of patients are progressing after initial response to checkpoint blockade immunotherapy. The field is undertaking major task to identify suitable combinatorial approach to improve the efficacy of checkpoint blockade immunotherapy and biomarker for better patient selection. Evidence suggests that EZH2 (Enhancer Zeste Homolog: enzymatic component of Polycomb Repressive Complex 2) plays a significant role in prognosis of patients with non-small cell lung cancer and animal studies showed that EZH2 targeting can improve the efficacy of immunotherapy.

Based on this, it was hypothesized that EZH2 inhibitor, tulmimetostat can re-sensitive cancer cells to respond to PD-1 blockade, pembrolizumab and designed phase Ib/II single arm, open label study to test this hypothesis for patients with advanced non-small cell lung cancer who progressed from front or second line of therapy (expecting majority of patients experienced checkpoint blockade immunotherapy). The primary objectives of this study are safety/tolerability and Objective Response Rate (ORR: Complete Response and Partial Response) evaluated by RECIST v1.1. Key secondary objectives are disease control rate, progression free survival at 1 year, and duration of response. The study will employ safety lead-in phase Ib using BOIN (Bayesian Optimal Interval Design) with 2 dose levels (200 and 300 mg) for tulmimetostat, starting 200mg mg orally once daily. Tulmimetostat will be administered for 7 days prior to pembrolizumab 200 mg intravenous every 3 weeks that is defined as run-in phase (only prior to first cycle). It is planned to enroll 18 patients during phase Ib to determine recommended dose for phase II (RP2D). The sample size for phase II was calculated using Simon optimum two-stage design in order to determine the futility at early time. In the first stage, 15 subjects will be enrolled. If 2 or more responses are observed, an additional 39 subjects will be accrued during second phase. If in total there are 8 or more responses, we will consider the drug combination worthy of further clinical development, provided other factors such as toxicity and progression-free survival also appear favorable. For this phase II portion, up to 54 subjects are enrolled. This design has a one-sided alpha of 5% and a power of 80%. Planned duration of enrollment is 2 years, correlative studies (methyl marker: H3K27me3 and PD-L1, exome, RNA, circulating ctDNA sequencing and immune monitoring) are proposed using tumor biopsies (on treatment biopsy is optional) and blood samples before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent/assent for the trial. The trial consent includes future biomedical research.
* Male/female participants who are at least 18 years of age on the day of signing informed consent
* Patients with histologically confirmed diagnosis of advanced non-small cell lung cancer.
* Have a life expectancy of 12 weeks
* Participants who progressed from chemo(platinum-based)-immunotherapy, immunotherapy single agent or immuno-immuno combination therapies as front or second line of therapy.
* Participants must have progressed on treatment with an anti-PD-1/L1 mAb administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria:

  1. Has received at least 2 doses of an approved anti-PD-1/L1 mAb.
  2. Has demonstrated disease progression after anti-PD-1/L1 as defined by RECIST v1.1. The initial evidence of PD is to be confirmed by a second assessment no less than 4 weeks from the date of the first documented disease progression, in the absence of rapid clinical progression (as defined in 4.c).
  3. Progressive disease has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb.

     1. Progressive disease is determined according to RECISTv1.1.
     2. This determination is made by the investigator. Once disease progression is confirmed, the initial date of disease progression documentation will be considered the date of disease progression.
* Have measurable disease per RECIST v1.1 as assessed by the investigator and site radiologist.
* Have provided archival tumor sample or newly obtained core or excisional biopsy of tumor lesion. Formalin fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides and the pretreatment biopsy is discretionary if suitable archival tissue sample is available.
* Adequate organ function. (must be within 10 days prior to start of study intervention)
* Absolute neutrophil counts (ANC) 1500/mm3
* Platelet count 100,000/mm3
* Hemoglobin 9 g/dL without need for hematopoietic growth factor or transfusion support.
* Serum creatinine 1.5 x ULN (Upper Limit of Normal), or 24-hour creatinine clearance 30 cc/min. (note: creatinine clearance need not be determined if the baseline serum creatinine is within normal limits)
* Serum bilirubin 1.5 ×ULN OR direct bilirubin ULN for participants with total bilirubin levels >1.5 × ULN.
* Aspartate amino transferase (AST) 2.5 ULN or 5XULN for subjects with liver metastases.
* Alanine amino transferase (ALT) 2.5 ULN or 5XULN for subjects with liver metastases.
* Alkaline phosphatase 2.5 X ULN of liver fraction if 2.5 X ULN
* Serum albumin 2.5g/dL.
* Prothrombin time (PT) 1.5 x ULN and INR 1.3
* Partial thromboplastin time (PTT) 1.5 ULN.
* ECOG 0-1.
* Allowing patients who received over 30 Gy radiation therapy within 6 months of pembrolizumab treatment given the safety data from stage III patient received immunotherapy after concurrent chemotherapy and radiation.
* Female subjects of childbearing/reproductive potential must have a negative serum pregnancy test within 72 hours prior to receiving the treatment of study medication.
* Female subjects of childbearing potential and their partners must be willing to use a highly effective method of contraception as outlined in 5.5.2- Contraception, for the course of study through 183 days after the last dose of study medication.
* Male subjects and their partners of childbearing potential must agree to use a highly effective method of contraception as outlined in 5.5.2- Contraception, starting with the first dose of study medication through 183 days after the last dose of therapy and refrain from donating sperm during this period.

Note: both for male and female subjects, abstinence is acceptable if this is life style or preferred method of contraception

Exclusion Criteria:

* Primary diagnosis of low to intermediate grade of neuroendocrine lung cancer.
* Clinically active cerebral metastases. Patients with a prior diagnosis of cerebral metastases may be enrolled, provided that lesions have been adequately treated with radiation therapy or surgery, and have not required steroids for at least one month prior to study initiation.
* Is currently participating in or has participated in a study of an investigational agent within 4 weeks prior to study enrollment.

Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

Note: Participants must have recovered from all AEs due to previous therapies to Grade 1 or baseline. Participants with Grade 2 neuropathy may be eligible. Participants with endocrine-related AEs Grade 2 requiring treatment or hormone replacement may be eligible

* Prior exposure to tulmimetostat or other EZH2 inhibitors.
* EGFR or ALK altered patients.
* Immunotherapy naïve patients.
* Has a history of severe hypersensitivity reaction to pembrolizumab ( Grade 3).
* Has an active autoimmune disease that requires systemic treatment within the past 2 years or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic immunosuppressive agents, such as more than 10 mg of prednisone per day to control the disease. Patients with vitiligo or resolved childhood asthma/atopy would be exception to this rule. Patient requiring intermittent use of bronchodilator or local steroid would not be excluded. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not excluded from the study.
* Patient is positive for Human Immunodeficiency Virus (HIV) (HIV 1 2 antibodies), active Hepatitis B (HBsAg reactive) or Hepatitis C (HCV RNA is detected); patients with negative Hepatitis C antibody testing may not need RNA testing.
* History of non-infectious pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has received a live virus vaccine or live-attenuated within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
* Subjects taking medications that are known as strong CYP3A4 inducers/inhibitors.

(examples of inducers: not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, and St. John's wort; examples of inhibitors: not limited to atazanavir, clarithromycin, indinavir, itraconazole, troleandomycin, voriconazole, and grapefruit or grapefruit juice. Please refer to this website for the full information: http://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/ DrugInteractionsLabeling/ucm080499.htm; http://medicine.iupui.edu/clinpharm/ddis/)

* Has not fully recovered from any effects of major surgery without significant detectable infection. Surgeries that required general anesthesia or major surgeries must be completed at least 4 weeks before first study intervention administration. Surgery requiring regional/epidural anesthesia must be completed at least 72 hours before first study intervention administration and participants should be recovered.
* Has received prior radiotherapy within 4 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation ( 2 weeks of radiotherapy) to non-CNS disease.
* Had administered concomitant medication(s) or food or beverage that are strong CYP3A inducers or inhibitors within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 year. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Inability to take oral medication or malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea, or vomiting) that might impair the bioavailability of tulmimetostat.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Venous thromboembolism or pulmonary embolism within the last 3 months before starting study medication.
* Subjects who undergone an allogenic tissue/solid organ transplantation.
* A WOCBP who has a positive serum pregnancy test within 72 hours prior to study treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Pregnant female subjects or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 183 days after the last dose of study treatment.
* Patient is, at the time of signing consent, current use of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol)
* Has known psychiatric disorders that would interfere with cooperation with the requirement of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-12-08 (Estimated); Study Completion 2029-12-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  ORR assessed by RECIST v1.1
Safety and Tolerability | 2 years
  Safety and tolerability assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Disease control rate (DCR) | 2 years
  DCR (complete response, partial response and stable disease) assessed by RECIST v1.1
Progression Free Survival (PFS) and 1-year survival rate | 1 year
  PFS assessed by Kaplan Meyer survival analysis.
Duration of Response (DOR) | 2 years
  DOR assessed by RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Shin, MD PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (5):
- United States (5):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Northern California Health Care System, Mather, CA, Sacramento, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: No